CLINICAL TRIAL: NCT00016198
Title: A Randomized, Multicenter, Phase II Study Of Bolus/Infusion 5-FU/LV (de Gramont Regimen) Versus Oxaliplatin And Bolus/Infusion 5-FU/LV (de Gramont Regimen) As Third-Line Treatment Of Patients With Metastatic Colorectal Carcinoma
Brief Title: Fluorouracil and Leucovorin With or Without Oxaliplatin in Treating Patients With Recurrent Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prologue Research International (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: PROLOGUE-EFC4760; CDR0000068606 (Registry Identifier: PDQ (Physician Data Query)); SANOFI-EFC4760
Record Dates: First submitted 2001-05-06; First posted 2004-01-07 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2010-12

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Folfox protocol; Fluorouracil; Leucovorin; Oxaliplatin

INTERVENTIONS:
Drug: FOLFOX regimen
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Randomized phase II trial to study the effectiveness of combining fluorouracil and leucovorin with or without oxaliplatin in treating patients who have recurrent metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the overall response rate and overall survival of patients with recurrent metastatic colorectal adenocarcinoma treated with third-line therapy comprising fluorouracil and leucovorin calcium with or without oxaliplatin. II. Compare the onset and duration of complete and partial responses and duration of disease stabilization in patients treated with these regimens. III. Compare the proportion of patients with stable disease and proportion of patients with tumor-related symptomatic improvement treated with these regimens. IV. Compare the time to disease progression and time to tumor-related symptomatic worsening in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms. Arm I: Patients receive leucovorin calcium IV over 2 hours and fluorouracil IV over 2-4 minutes followed by fluorouracil IV continuously over 22 hours on days 1 and 2. Arm II: Patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV over 2-4 minutes followed by fluorouracil IV continuously over 22 hours on day 1. On day 2, patients receive leucovorin calcium and fluorouracil as in arm I. Treatment in both arms repeats every 2 weeks for at least 1 year in the absence of disease progression. Patients are followed at day 30 and then for approximately 6 months.

PROJECTED ACCRUAL: A total of 200 patients (100 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed adenocarcinoma of the colon or rectum Metastatic/recurrent disease not amenable to potentially curative therapy (e.g., inoperable metastatic disease) Documented sequential disease progression (by CT scan or MRI) after 2 prior chemotherapy regimens for metastatic/recurrent disease At least 1 unidimensionally measurable lesion At least 20 mm by conventional CT scan or MRI OR At least 10 mm by spiral CT scan Must have received prior fluorouracil (or capecitabine) and leucovorin calcium with or without irinotecan as first-line therapy and irinotecan with or without fluorouracil (or capecitabine) and leucovorin calcium as second-line therapy for metastatic disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 50-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT and SGPT no greater than 2 times ULN (6 times ULN if documented liver metastases present) Alkaline phosphatase no greater than 2 times ULN (6 times ULN if documented liver metastases present) Renal: Creatinine no greater than 1.5 times ULN Cardiovascular: No New York Heart Association class III or IV symptomatic congestive heart failure No serious cardiac arrhythmia No unstable angina No myocardial infarction within the past 6 months Pulmonary: No interstitial pneumonia No extensive and symptomatic fibrosis of the lung Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 6 months after study No known peripheral neuropathy (absence of deep tendon reflexes as the sole neurologic abnormality allowed) No diabetes or active infection No known dihydropyrimidine dehydrogenase deficiency

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior anticancer biologic therapy Chemotherapy: See Disease Characteristics No prior oxaliplatin No prior adjuvant irinotecan Prior adjuvant fluorouracil and leucovorin calcium allowed At least 3 weeks since prior chemotherapy (e.g., second-line irinotecan with or without fluorouracil (or capecitabine) and leucovorin calcium) for metastatic disease and recovered Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since prior radiotherapy No prior radiotherapy to target lesion unless documented progression within the radiation portal Surgery: See Disease Characteristics At least 4 weeks since prior surgery for primary tumor or metastases and recovered Other: No prior investigational anticancer drug No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-05; Primary Completion 2003-04 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Gams, MD, Study Chair — Prologue Research International
Locations (74):
- United States (74):
  - Arizona Clinical Research Center, Tucson, Arizona
  - Arkansas Cancer Clinic, P.A., Pine Bluff, Arkansas
  - Citrus Valley Medical Center, Covina, California
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - California Cancer Care, Inc., Greenbrae, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Kenmar Research Institute, Los Angeles, California
  - Comprehensive Cancer Centers of the Desert, Palm Springs, California
  - Kaiser Permanente-Southern California Permanente Medical Group, San Diego, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - John Muir Medical Center, Walnut Creek, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Northwestern Connecticut Oncology-Hematology Associates, Torrington, Connecticut
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Center for Hematology-Oncology, Boca Raton, Florida
  - Halifax Medical Center, Daytona Beach, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Hematology/Oncology Associates, Jacksonville, Florida
  - Lake Heart and Cancer Medical Center, Leesburg, Florida
  - Oncology-Hematology Group of South Florida, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Hematology/Oncology Associates, Port Saint Lucie, Florida
  - Northwest Medical Specialists, P.C., Arlington Heights, Illinois
  - Dreyer Medical Clinic, Aurora, Illinois
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, S.C., Decatur, Illinois
  - Hope Center, Terre Haute, Indiana
  - Medical Oncology and Hematology Associates, Des Moines, Iowa
  - Mercy Cancer Center, Mason City, Iowa
  - Lucille Parker Markey Cancer Center, University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Cancer and Blood Institute, Metairie, Louisiana
  - Saints Memorial Medical Center, Lowell, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Medical Oncology Group, Gulfport, Mississippi
  - Jackson Oncology Associates, PLLC, Jackson, Mississippi
  - St. Joseph Oncology, Inc., Saint Joseph, Missouri
  - Deaconess Billings Clinic, Billings, Montana
  - Monmouth Medical Center, Long Branch, New Jersey
  - Jersey Shore Cancer Center, Neptune City, New Jersey
  - Central Jersey Oncology Center, New Brunswick, New Jersey
  - Hematology Associates of New Jersey, P.A., Ridgewood, New Jersey
  - Monmouth Hematology-Oncology Associates, P.A., West Long Branch, New Jersey
  - University of New Mexico Cancer Research & Treatment Center, Albuquerque, New Mexico
  - HemOnCare, P.C., Brooklyn, New York
  - North Shore Hematology/Oncology Associates, P.C., East Setauket, New York
  - Reddy Cancer Treatment Center, Malone, New York
  - New York University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - South Shore Hematology Oncology Associates, P.C., Rockville Centre, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mid-Ohio Oncology/Hematology, Inc., Columbus, Ohio
  - Hematology Oncology Consultants Inc, Columbus, Ohio
  - Lawrence M. Stallings Medical Practice, Wooster, Ohio
  - Oklahoma Oncology Inc., Tulsa, Oklahoma
  - Bend Memorial Clinic, Bend, Oregon
  - Salem Hospital Regional Cancer Center, Salem, Oregon
  - Oncology Hematology of Lehigh Valley, P.C., Bethlehem, Pennsylvania
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Memorial Hospital Cancer Center - Chattanooga, Chattanooga, Tennessee
  - Family Cancer Center, Collierville, Tennessee
  - Baptist Regional Cancer Center, Knoxville, Tennessee
  - West Cancer Clinic, Memphis, Tennessee
  - Center for Oncology Research and Treatment, Medical City Hospital, Dallas, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Intermountain Hematology/Oncology Associates, Inc., Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington